CLINICAL TRIAL: NCT05234398
Title: TIXAGEVIMAB/CILGAVIMAB for Covid-19 Pre-exposition Prophylaxis in Solid Organ Transplanted Recipients
Brief Title: TIXAGEVIMAB/CILGAVIMAB Protection of Covid-19 in Transplanted Patients
Acronym: TIXCI-TRANS
Status: Withdrawn | Type: Observational
Why Stopped: This project will be integrated into an ongoing project.
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: 69HCL21_1433; 2021-A03245-36 (Other: ID-RCB)
Record Dates: First submitted 2022-02-08; First posted 2022-02-10 (Actual); Last update posted 2022-09-01 (Actual); Status verified 2022-08

CONDITIONS: Solid Organ Transplant Recipients
Keywords: monoclonal antibody; protective level of SARS CoV2 antibodies; pharmacokinetic of anti-SARS CoV2 antibodies; SARS CoV2 infection; viral neutralization capacity; anti-Nucleocapsid IgG (Immunoglobulin G)
MeSH Terms: conditions — COVID-19 | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Naïve patients: This study involve non-responder solid organ transplanted patients after an adapted vaccinal scheme (i.e. 3 doses or more of mRNA vaccines).
  Patients included in Group 1 are naïve patients; there have never received anti-SARS Cov2 monoclonal antibodies.
  They will have additional blood and saliva samplings during their study visits, which are included in their usual medical follow-up.
  Interventions: Biological: Blood and saliva samplings
- Switched patients: This study involve non-responder solid organ transplanted patients after an adapted vaccinal scheme (i.e. 3 doses or more of mRNA vaccines).
  Patients included in Group 2 have previously received anti-SARS Cov2 monoclonal antibodies.
  They will have additional blood and saliva samplings during their study visits, which are included in their usual medical follow-up.
  Interventions: Biological: Blood and saliva samplings

INTERVENTIONS:
Biological: Blood and saliva samplings — At each protocol visits, on the occasion of a care collection, additional blood and saliva samples will be taken specifically for the study, with a total volume of blood of 38 mL, and a saliva sample of 1.5 to 2 mL per visit (inclusion, month 1, month 4, month 6, month 9 and month 12), corresponding to routine care.

SUMMARY:
Covid-19 has a very bad prognosis in solid organ transplant recipients with a 60 days-mortality exceeding 20%. For this reason, transplant patients were prioritized to receive Covid-19 vaccination since December 2020 in France. Unfortunately, the vaccine response of these patients is insufficient after a standard vaccine regimen including 2 doses of mRNA (messenger ribonucleic acid) vaccine with a 50% seroconversion rate in many cohorts. As a result, on the advice of the "Conseil National d'Orientation Vaccinale", the French Health Authorities has authorized physicians to offer a 3rd dose of vaccine to organ transplant patients since April 11, 2021. The subsequent studies showed that half of the patients who did not seroconvert after the 2nd dose did develop a vaccine response after the third dose. For patients who do not respond after the 3rd dose, the clinicians are now allowed to offer a 4th dose of vaccine.

Unfortunately, approximately 25% of patients still remain non-responders to this 3- or 4-doses vaccine regimen. In addition, transplant recipients who do not developed a vaccine response after the 3rd dose are very unlikely to respond after the 4th dose. For patients who do not respond to the vaccination, the French Health Authorities had authorized the infusion of SARS Cov2 (Severe Acute Respiratory Syndrome Coronavirus 2) monoclonal antibodies as a pre-exposition prophylaxis in immunocompromised patients.

The value of using the TIXAGEVIMAB/CILGAVIMAB monoclonal antibody cocktail as primary prophylaxis has been demonstrated in the general population but this study did not include immunocompromised patients.

Here, the investigators propose to study the pharmacokinetics of TIXAGEVIMAB/CILGAVIMAB given in a pre-exposition prophylaxis scheme in non-responder solid organ transplanted patients after an adapted vaccinal scheme (i.e. 3 doses or more of mRNA vaccines).

ELIGIBILITY:
Inclusion Criteria:

* Male or female, 18 years of age or older
* Recipient of a solid organ transplant
* Subject affiliated with a health insurance company
* Patient able to understand the objectives and risks of the research and to give a non-objection
* Patient with a post-vaccination anti-Spike IgG (or RBD - Receptor Blinding Domain) titer of less than 30 BAU/ml ( (binding antibody units) measured at least 14 days after completion of an intensified vaccination regimen (at least 3 doses of mRNA vaccine) and prior to administration of anti-SARS-Cov-2 monoclonal antibodies.
* Group 1 criteria: Naïve patients, never having received anti-SARS CoV2 monoclonal antibodies.
* Group 2 criteria: Patients who have previously received anti-SARS Cov2 monoclonal antibodies

Exclusion Criteria:

* History of anaphylactic shock or known allergy to TIXAGEVIMAB/CILGAVIMAB
* Known history of Covid-19 or positive Covid-19 serology within 3 months prior to inclusion
* History of myocardial infarction or coronary artery disease within 3 months prior to inclusion
* Contraindication to an intramuscular injection
* Impossibility to give to the subject an informed information
* Subject under legal protection, guardianship or curatorship
* Plasmapheresis in progress or planned
* Weight less than 48 kg
* Patient participating in another interventional research study in progress
* Pregnant, parturient, or breastfeeding women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 160 solid organ transplant patients will be enrolled in the study. Recruitment will be performed among transplant patients at the two transplant centers participating in the study during a follow-up visit, after receipt of their serology results.
  Patients will be allocated into two groups:
  * Group 1 (100 patients): naïve patients, who have never received anti-SARS CoV2 monoclonal antibodies.
  * Group 2 (60 patients): patients who have previously received anti-SARS Cov2 monoclonal antibodies.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2022-02 (Estimated); Primary Completion 2023-02 (Estimated); Study Completion 2023-08 (Estimated)

PRIMARY OUTCOMES:
Percentage of patients whose serum has viral neutralization capacity in vitro at M6 after TIXAGEVIMAB/CILGAVIMAB injection. | At Month 6.
  Viral neutralization capacity will be analyzed by performing in-vitro neutralization tests from blood samples of enrolled patients.
  Samples will be analyzed centrally by virology Laboratory of Strasbourg Hospital throughout the study.

CONTACTS AND LOCATIONS:
Overall Officials: Olivier THAUNAT, MD-PhD, Principal Investigator — Service de Néphrologie, Transplantation et Immunologie Clinique Hôpital Edouard Herriot - Hospices Civils de Lyon
Locations (2):
- France (2):
  - Service de Néphrologie, Transplantation et Immunologie Clinique Hôpital Edouard Herriot - Hospices Civils de Lyon, Lyon
  - Service de Néphrologie et Transplantation, Hôpitaux Universitaires de Strasbourg, Strasbourg